CLINICAL TRIAL: NCT03616717
Title: Neurophysiological Biomarkers of Behavioral Dimensions From Cross-species Paradigms
Brief Title: Modafinil Effects on EEG Biomarkers of Reward and Motivation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jared W. Young, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 4UH3MH109168-03 (NIH)
Record Dates: First submitted 2018-07-18; First posted 2018-08-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Modafinil

STUDY DESIGN:
Intervention Model Description: Experimental medicine model; not an intervention. Within-subject double-blind placebo-controlled dose-response study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: University of California, San Diego Experimental Pharmacy randomizes dose order and provides masked pills
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- modafinil 100 mg (Active Comparator): Drug: modafinil, Provigil, Alertec, Modavigil
  Dosage form, frequency and duration: Each participant receives a single pill of placebo or active drug (modafinil 100 mg or 200 mg) 30 minutes after arriving at the lab. The participant then completes approximately 6 hours of testing in the laboratory. The participant stays at the lab for 7.5 hours in order to monitor physical condition in case the participant received the active pill. One week later, that participant receives a single pill of an alternate comparator and is again tested in the laboratory. Thus, in total, each participant receives one placebo pill and two active pills, each time separated by one week.
  Interventions: Drug: Modafinil
- modafinil 200 mg (Active Comparator): Drug: modafinil, Provigil, Alertec, Modavigil
  Dosage form, frequency and duration: Each participant receives a single pill of placebo or active drug (modafinil 100 mg or 200 mg) 30 minutes after arriving at the lab. The participant then completes approximately 6 hours of testing in the laboratory. The participant stays at the lab for 7.5 hours in order to monitor physical condition in case the participant received the active pill. One week later, that participant receives a single pill of an alternate comparator and is again tested in the laboratory. Thus, in total, each participant receives one placebo pill and two active pills, each time separated by one week.
  Interventions: Drug: Modafinil
- placebo (Placebo Comparator): Drug: modafinil, Provigil, Alertec, Modavigil
  Dosage form, frequency and duration: Each participant receives a single pill of placebo or active drug (modafinil 100 mg or 200 mg) 30 minutes after arriving at the lab. The participant then completes approximately 6 hours of testing in the laboratory. The participant stays at the lab for 7.5 hours in order to monitor physical condition in case the participant received the active pill. One week later, that participant receives a single pill of an alternate comparator and is again tested in the laboratory. Thus, in total, each participant receives one placebo pill and two active pills, each time separated by one week.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Modafinil — Drug: modafinil Each participant receives a single pill of placebo or active drug (modafinil 100 mg or 200 mg) 30 minutes after arriving at the lab. The participant then completes approximately 6 hours of testing in the laboratory. The participant stays at the lab for 7.5 hours in order to monitor physical condition in case the participant received the active pill. One week later, that participant receives a single pill of an alternate comparator and is again tested in the laboratory. Thus, in total, each participant receives one placebo pill and two active pills, each time separated by one week.
  Other Names:
  Provigil Alertec Modavigil
  Arms: modafinil 100 mg; modafinil 200 mg
Drug: placebo — Drug: Placebo Each participant receives a single pill of placebo or active drug (modafinil 100 mg or 200 mg) 30 minutes after arriving at the lab. The participant then completes approximately 6 hours of testing in the laboratory. The participant stays at the lab for 7.5 hours in order to monitor physical condition in case the participant received the active pill. One week later, that participant receives a single pill of an alternate comparator and is again tested in the laboratory. Thus, in total, each participant receives one placebo pill and two active pills, each time separated by one week.
  Arms: placebo

SUMMARY:
The effects of modafinil on measures of brain electrical activity will be tested.

ELIGIBILITY:
Exclusion criteria

* history of substance abuse
* mental illness in a first degree relative
* significant medical illness (e.g. cancer, diabetes, heart disease, HIV)
* history of seizure
* open head injury or closed head injury with loss of consciousness > 1 min
* pregnancy
* current psychotropic drug use
* R-hand injury
* hearing or visual impairment
* urine toxicology positive for recreational drug use

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Reward Positivity | 1 year
  Frontal alpha power by block in the probabilistic learning task
Motivation Signal | 1 year
  Parietal EEG alpha power peak in first - final step toward breakpoint

CONTACTS AND LOCATIONS:
Overall Officials: Jared W Young, Ph.D., Principal Investigator — UCSD
Locations (1):
- University of California, San Diego; Clinical Teaching Facilities, Hillcrest, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No